CLINICAL TRIAL: NCT06189807
Title: Pregnancy and Contraception Education in Chronic Kidney Disease (PACE-CKD): A Pilot Study
Brief Title: Pregnancy and Contraception Education in Chronic Kidney Disease (PACE-CKD)
Acronym: PACE-CKD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Andrea Oliverio, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00233787; 1K23DK123413-01A1 (NIH)
Record Dates: First submitted 2023-12-18; First posted 2024-01-05 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: CKD; Chronic Kidney Diseases
Keywords: Pregnancy and Contraception education
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Decision Support Techniques

STUDY DESIGN:
Intervention Model Description: Group assignment will be randomized at the clinic level to intervention decision aid (N=2 clinics) or control (N=2 clinics). Nephrologists will be trained to deliver the intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group - (Other)
  Interventions: Other: Standard handout
- Intervention Group - Decision aid (Experimental)
  Interventions: Behavioral: Decision aid

INTERVENTIONS:
Behavioral: Decision aid — Enrolled participants will be sent the novel educational decision aid about pregnancy, birth control, and kidney disease and asked to read that information prior to a standard of care appointment with participants nephrologist. Prior to the appointment, study staff will provide participants with a paper version of the materials that had previously been sent. During the appointment participant's nephrologist may review the materials with the participant and answer any questions. Following the appointment, participants will be asked to complete a short survey about: the experience using the materials, experience about being counseled about pregnancy and birth control during visit, willingness to use such materials in the future, and information about participants kidney disease diagnosis.
  Arms: Intervention Group - Decision aid
Other: Standard handout — Enrolled participants will be sent the standard information about pregnancy, birth control, and kidney disease and asked to read that information prior to a standard of care appointment with participants nephrologist. Prior to the appointment study staff will provide participants with a paper version of the materials that had previously been sent. During the appointment, the participant's nephrologist may review the materials with the participant and answer any questions. Following the appointment, participants will be asked to complete a short survey about: the experience using the materials, experience about being counseled about pregnancy and birth control during visit, willingness to use such materials in the future, and information about participants kidney disease diagnosis.
  Arms: Control Group -

SUMMARY:
This pilot study will assess the efficacy of a pregnancy and contraception education decision aid (DA) for patients with chronic kidney disease to support decisions about reproductive health, and will assess feasibility and acceptability of the intervention to inform future Research Project Grant (R01) level studies.

DETAILED DESCRIPTION:
60 patient participants will receive either a novel DA about pregnancy and contraception in chronic kidney disease delivered by patient's nephrologist or will receive currently available educational materials based on clinic-level randomization. Nephrologists will be trained to deliver the novel decision aid or will provide usual care. Patients will complete a survey about pregnancy and contraception decision making and the acceptability and feasibility of the educational materials after the clinical visit. Intervention nephrologists will be anonymously surveyed after all patients have completed measures, to assess acceptability and feasibility.

ELIGIBILITY:
Inclusion Criteria:

* Any Chronic Kidney Disease (CKD) diagnosis
* CKD defined as abnormality in kidney structure or function for >3 months and may be manifested by having any one of the following:

  i. Glomerular filtration rate (GFR)<60 milliliter/Minute (ml/min)/1.73m2, or

ii. A marker of kidney damage (albuminuria >30 milligrams per gram (mg/g), abnormal kidney histology by biopsy, hematuria, structural abnormalities by imaging (e.g. polycystic kidney disease, horseshoe kidney) or electrolyte abnormalities due to tubular disorders)

- Able to speak and read English

Exclusion Criteria:

* Patients receiving dialysis
* Patients who have a kidney transplant
* Patients that are surgically sterile (tubal ligation or hysterectomy) or currently pregnant
* Patients that have significant cognitive or visual impairment that limits interaction with the decision aid (DA)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-02-14 (Actual); Primary Completion 2025-09-24 (Actual); Study Completion 2026-09-25 (Estimated)

PRIMARY OUTCOMES:
Preparation for Decision Making (PrepDM) score at post-intervention | Day 1- 7 (post appointment with provider)
  This is a 10-item survey that participants answer not at all (1) to a great deal (5).
  PrepDM is scored on a 0-100 scale, where higher score indicates better preparation for decision making. A score of >75 is a clinically significant cut off that indicates participants being well prepared to make decisions after reviewing a DA.The PrepDM scale was adapted slightly to meet the needs of the target population and the developed novel decision aid.

SECONDARY OUTCOMES:
Feasibility of delivering a reproductive health decision aid in an academic nephrology clinic measured by proportion of approached patients that consent during screening period | 12 months (after recruitment starts)
Feasibility of delivering a reproductive health decision aid in an academic nephrology clinic measured by the percentage of enrolled patients in the intervention clinics that providers reviewed contraception or pregnancy planning with participants during | Day 1 (Visit at the clinic)
Acceptability of delivering a reproductive health decision aid in a nephrology clinic -participants | Day 1- 7 (post appointment with provider)
  Acceptability of using the shared decision aid will be assessed by 8 questions and analyzed descriptively.
Acceptability of delivering a reproductive health decision aid in a nephrology clinic- nephrologists | 12 months
  Acceptability of using the shared decision aid will be assessed by 2 questions and analyzed descriptively.
Feasibility of delivering a reproductive health decision aid in a nephrology clinic - nephrologists | 12 months
  Feasibility of using the shared decision aid will be assessed by 2 questions and analyzed descriptively.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Oliverio, MD, MSc, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-03-20): https://cdn.clinicaltrials.gov/large-docs/07/NCT06189807/ICF_000.pdf